CLINICAL TRIAL: NCT07183644
Title: Maximizing Laser Therapy Success for Port-Wine Birthmarks in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James Seaward, Board Certified Plastic Surgeon, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stu-2024-1203
Record Dates: First submitted 2025-09-07; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Port Wine Stains
Keywords: combined laser therapy; PDL; Nd:YAG laser; port wine stain; port wine birthmark
MeSH Terms: conditions — Hemangioma, Capillary; Port-Wine Stain | interventions — Lasers, Solid-State; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All patients (Active Comparator): Every patient will receive the 5 treatment modalities in their first laser treatment after enrollment in the study.
  * At 5-7 weeks follow-up visit after the procedure, if no treatment modality is better than the other, then the surgeon will repeat the procedure with the 5 modalities, and the subject will have a 2nd follow-up appointment 5-7 weeks later. Continue treatment with 5 modalities and appropriate follow-up until Port Wine Birthmark (PWB) clearance, or,
  * If any modality is seen to give best results at the first follow-up visit (5-7 weeks after the first procedure), then the next treatment will be only with that modality and will continue to have treatments with this modality and follow-up appointments (5-7 weeks after procedure) according to standard of care timelines for PWBs until the treatment is not improving the PWB anymore or until the PWB is no longer visible.
  Interventions: Device: Pulse Dye laser; Device: Pulse Dye Laser (PDL) pulse width stacking; Device: Pulse Dye Laser (PDL) followed by Nd:YAG (Neodymium-doped Yttrium Aluminum Garnet laser) laser.; Device: IPL (Intense Pulsed Light) followed by Pulse Dye Laser (PDL); Device: Cupping followed by Pulse Dye Laser (PDL)

INTERVENTIONS:
Device: Pulse Dye laser — Pulse Dye Laser (PDL) standard settings. This is the same procedure children would receive as standard of care if these individuals were not participating in this study.
  The surgeon will perform 1 pass with the PDL over the area of the Port wine birthmark (PWB).
Device: Pulse Dye Laser (PDL) pulse width stacking — This procedure is used for some patients as standard of care depending on the severity and depth of the lesion.
  The surgeon will perform 3 passes with the PDL over the PWB, gradually increasing the pulse duration with each pass to effectively target both superficial and deeper blood vessels.
Device: Pulse Dye Laser (PDL) followed by Nd:YAG (Neodymium-doped Yttrium Aluminum Garnet laser) laser. — The combination of these two lasers is one of the investigational treatments. The surgeon will perform 1 pass per laser over the PWB. The 1st pass will be with the PDL to target the blood vessels closer to the top of the skin, followed by a 2nd pass with the Nd:YAG laser to target the blood vessels that deeper in the skin.
Device: IPL (Intense Pulsed Light) followed by Pulse Dye Laser (PDL) — The surgeon will perform 1 pass with the IPL followed by 1 pass with the PDL over the PWB
Device: Cupping followed by Pulse Dye Laser (PDL) — The combination of these modalities is one of the experimental procedures. The surgeon will place a small suction cup over the PWB target region of the PDL for a few seconds to stop the blood flow and accumulate the blood in that spot. The PDL treatment will then quickly proceed. Since the PDL targets red blood cells, it will allow the laser to target the pooled blood in the abnormal blood vessels better.

SUMMARY:
In this study the investigators aim to optimize Port-Wine-Birthmark (PBW) laser therapy in children in order to reduce the number of laser treatments required for clearance and improve outcomes for refractory cases. This approach also seeks to reduce the frequency with which children require general anesthesia for treatment.

DETAILED DESCRIPTION:
Participants will undergo up to two laser treatment sessions on the Port-Wine Birthmark (PWB), in which five treatment modalities will be applied. The modality with the best outcomes will be used for subsequent treatments until the PWB is cleared or treatment with that modality reaches an outcome plateau, as determined by the treating physician. If no further outcome response is observed with that modality, the patient will undergo a second round of the five different modalities to determine if there are differences in efficacy. The treatment modality showing the best response will then be continued. Patient outcomes will then be analyzed to determine if there are significant differences between treatment modalities as well as among primary treatment patients and refractory cases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Port Wine Stain.
* Age Range: 2mo to 18 years of age.
* Stable PWS: The port wine stain should be stable, meaning there is no active inflammation or infection present, and it should not be changing in size or color due to factors like injury or disease.
* signed Consent: For ethical reasons, participants must be able to provide informed consent. In the case of minors, consent would generally be required from a parent or legal guardian.

General Health: Participants should generally be in good health, with no contraindications for laser therapy, such as certain skin conditions, infections, or hypersensitivity to light.

Exclusion Criteria:

* severe allergies to anesthesia
* active skin infections or inflammation
* recent laser therapy
* use of Photosensitizing medications
* participation in other laser studies

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Port Wine Birthmark (PWB) color in participants - Pre Operative | Baseline
  Prior to treatment, the PWB will be documented photographically. Images taken will be transformed in to the L a*b* colorspace (also known as the red green color axis), and regions of interest defined on the photographs corresponding with the areas treated by each modality, as well as a region of interest adjacent to the treated area, to act as a control to correct for skin changes unrelated to the treatment. The axis is representative of color chromaticity and is measured in a range of -128 to 127. Positive values are indicative of red, and negative values are indicative of green.
  The quantitative values of the a* channel in the L a*b* colorspace will be used as a measure of the PWB intensity and each treated area will be compared with the corresponding area pre-treatment, using the difference in a* values to determine the treatment effectiveness.
Change in Port Wine Birthmark (PWB) color in participants - Post Operative | 6 weeks
  Post-operatively, the treated area will once more be documented photographically.
  Images taken will be transformed in to the L a*b* colorspace (also known as the red green color axis), and regions of interest defined on the photographs corresponding with the areas treated by each modality, as well as a region of interest adjacent to the treated area, to act as a control to correct for skin changes unrelated to the treatment. The axis is representative of color chromaticity and is measured in a range of -128 to 127. Positive values are indicative of red, and negative values are indicative of green.
  The quantitative values of the a* channel in the L a*b* colorspace will be used as a measure of the PWB intensity and each treated area will be compared with the corresponding area pre-treatment, using the difference in a* values to determine the treatment effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: James Seaward, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Children's Medical Center, Dallas, Texas
  - Children's Medical Center, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
We will share the information based on the results of our study and a careful assessment of its potential value in treating this condition. Our decision will consider how the findings contribute to advancing knowledge and improving patient care.

REFERENCES:
- [Background] Chen JK, Ghasri P, Aguilar G, van Drooge AM, Wolkerstorfer A, Kelly KM, Heger M. An overview of clinical and experimental treatment modalities for port wine stains. J Am Acad Dermatol. 2012 Aug;67(2):289-304. doi: 10.1016/j.jaad.2011.11.938. Epub 2012 Feb 3. PMID 22305042
- [Background] Jasim ZF, Handley JM. Treatment of pulsed dye laser-resistant port wine stain birthmarks. J Am Acad Dermatol. 2007 Oct;57(4):677-82. doi: 10.1016/j.jaad.2007.01.019. Epub 2007 Jul 19. PMID 17658196
- [Background] Lee JW, Chung HY. Capillary Malformations (Portwine Stains) of the Head and Neck: Natural History, Investigations, Laser, and Surgical Management. Otolaryngol Clin North Am. 2018 Feb;51(1):197-211. doi: 10.1016/j.otc.2017.09.004. PMID 29217063
- [Background] Ahcan U, Zorman P, Recek D, Ralca S, Majaron B. Port wine stain treatment with a dual-wavelength Nd:Yag laser and cryogen spray cooling: a pilot study. Lasers Surg Med. 2004;34(2):164-7. doi: 10.1002/lsm.10252. PMID 15004829
- [Background] Li G, Lin T, Wu Q, Zhou Z, Gold MH. Clinical analysis of port wine stains treated by intense pulsed light. J Cosmet Laser Ther. 2010 Feb;12(1):2-6. doi: 10.3109/14764170903449778. PMID 20085450